CLINICAL TRIAL: NCT03274947
Title: An Exploration of the Application of Non-invasive Cerebellar Stimulation in the Neurorehabilitation of Dysphagia After Stroke
Brief Title: The Utility of Cerebellar Transcranial Magnetic Stimulation in the Neurorehabilitation of Dysphagia After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Medical Research Council (Other Government); University of Nottingham (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5111 protocol ver1
Record Dates: First submitted 2017-08-14; First posted 2017-09-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Oropharyngeal Dysphagia; Stroke
Keywords: Oropharyngeal Dysphagia; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Hypothesis 2 Protocol 2 Low dose TMS (Active Comparator): Low level cerebellar TMS. Delivered once per day for 3 days.
  Interventions: Device: Cerebellar TMS
- Hypothesis 2 Protocol 2 High dose TMS (Active Comparator): High level cerebellar TMS. Delivered twice per day for 5 days.
  Interventions: Device: Cerebellar TMS
- Hypothesis 2 Protocol 2 Sham (Sham Comparator): Sham cerebellar TMS. Delivered twice a day for 5 days.
  Interventions: Device: Sham cerebellar TMS
- Hypothesis 2 Protocol 1 Cerebellar TMS (Active Comparator): Cerebellar TMS at 10Hz, 250 pulses.
  Interventions: Device: Cerebellar TMS
- Hypothesis 2 Protocol 1 Sham (Sham Comparator): Sham cerebellar TMS
  Interventions: Device: Sham cerebellar TMS

INTERVENTIONS:
Device: Cerebellar TMS — Cerebellar transcranial magnetic stimulation
  Arms: Hypothesis 2 Protocol 1 Cerebellar TMS; Hypothesis 2 Protocol 2 High dose TMS; Hypothesis 2 Protocol 2 Low dose TMS
Device: Sham cerebellar TMS — Sham cerebellar transcranial magnetic stimulation
  Arms: Hypothesis 2 Protocol 1 Sham; Hypothesis 2 Protocol 2 Sham

SUMMARY:
The study is designed to explore the effectiveness of non-invasive cerebellar stimulation to enhance motor plasticity in the cortex after stroke. The investigators have shown that the human cerebellum is strongly activated during the act of swallowing and when stimulated with single TMS pulses can strongly facilitate the corticobulbar projection to the pharynx in humans. More recently the investigators have identified the most relevant frequency of stimulation of the cerebellum that can produce longer term excitation in the human swallowing motor system. The investigators therefore believe that the potential for cerebellar stimulation in improving swallowing is much greater than other methods for two reasons. Firstly, previous work has shown that unlike successful recovery of hand/arm function which relies on restoring activity in the stroke hemisphere, recovery of swallowing function relies on increased excitability in intact projections from the non-stroke hemisphere. The investigators believe that methods that can enhance these undamaged pathways have a greater chance of inducing recovery in the human swallowing system in unilateral stroke. Additionally cerebellar stimulation produces very high levels of corticobulbar excitation it may also have the advantage of improving dysphagia in posterior fossa strokes. Second, the human cerebellum is relatively easy to target and stimulate and has reduced risk of inducing unwanted effects (such as seizures) which as a consequence makes cerebellar stimulation a more pragmatic method for delivering therapeutic neurorehabilitation to dysphagic stroke patients compared to other more complex/riskier methods.

A final factor is that the investigators have developed a "virtual lesion" model of swallowing dysfunction in healthy volunteers which can be reversed quite successfully with other neuro-stimulation protocols. The investigators can therefore use this model to test the effectiveness of cerebellar stimulation protocols (ipsilateral and contralateral cerebellar sites) before choosing the most effective side to apply stimulation in a proof of principle trial/study in a small group of sub-acute dysphagic patients.

The hypotheses are that cerebellar TMS will:

i. Reverse the brain inhibition and behavioural dysfunction following a virtual lesion model of disrupted swallowing in healthy brain (phase 1); ii. Reduce the degree of aspiration in acute dysphagia after a stroke (phase 2).

DETAILED DESCRIPTION:
Protocols:

Hypothesis 1:

Cortical excitability (in both dominant and non-dominant swallowing cortex) to TMS and swallowing behaviour assessed with a swallowing reaction time task will be measured at baseline. Thereafter, the virtual lesion paradigm will be applied to the dominant swallowing projection followed by the cerebellar intervention (10Hz, 250 pulses). Cerebellar stimulation will be applied (in a randomised fashion) on separate occasions to both the contralateral and ipsilateral cerebellar hemispheres, immediately after the virtual lesion. The investigators have found that placement using known reference landmarks are equivalent to using neuronavigation, so the latter will not be employed. Repeat measurements of cortical excitability and swallowing behaviour will then be performed and analysed against baseline data and a sham cerebellar paradigm. Differences in cortical excitability and swallowing responses will thus be an indication of which cerebellar region (contralesional/ipsilesional) can influence excitability and reverse any behavioural changes most effectively.

Hypothesis 2:

I. Dysphagic stroke patients (n=24) recruited over a 9 month period within 14 days of stroke ictus will have their swallowing assessed by videofluoroscopy before and after receiving either the real or sham cerebellar stimulation (10Hz, 250 pulses) as determined from phase 1. As before, placement of the coil for cerebellar stimulation will be performed using landmarks already established and validated in the work from question 1. Patients will be intubated with the pharyngeal EMG catheter for pre and post recordings of pharyngeal motor evoked potentials (MEPs) to cortical TMS. Power calculations, based on a similar study of pharyngeal stimulation indicated that the investigators would need 12 patients per group to achieve a statistical power of 80% at a 5% significance level to detect changes in the primary outcome measure of aspiration. In this study, the investigators will examine if the chosen site of cerebellar stimulation from phase 1 can induce short-term changes in brain function (pharyngeal MEPs) and swallowing function (videofluoroscopy) compared to sham interventions and baseline measurement, up to 1 hour after the intervention.

II. Following stage I, once it is established that cerebellar stimulation can alter brain and swallowing functions in stroke in the short-term, it will need to be appraised for clinical feasibility, dose response, and longer term efficacy. Dysphagic stroke patients (n=48, 16 patients per group) admitted to the stroke unit and identified by videofluoroscopy will be recruited over the next 21 months. Since it is not known how the cerebellar stimulation method should be delivered to patients, a dose ranging treatment trial will be utilised, randomising patients to one of three groups (A-C), low level stimulation, high level stimulation and sham stimulation. From our previous work with pharyngeal stimulation, the investigators propose that group A will receive stimulation once per day for 3 days. Group B will receive stimulation twice per day for 5 days. Group C will receive sham stimulation (delivered as in protocol I) twice a day for 5 days. Groups A and B will receive stimulation at the optimal site (10Hz, 250 pulses) found in question 1, but all groups will also receive standard speech and language therapy.

Assessments:

Swallowing before and after stimulation will be evaluated using videofluoroscopy, at 1 hour for protocol I. For protocol II the investigators propose both videofluoroscopy and functional scores (Functional oral ingestion scale (FOIS), the dysphagia severity rating scale (DSRS) including feeding status and modified rankin scale (mRS)) at baseline and at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* All patients with an acute anterior or posterior cerebral circulation stroke within 6 weeks of symptom onset.

Exclusion Criteria:

* Advanced dementia
* Previous history of dysphagia
* Patients judged to be clinically unstable
* Presence of implanted cardiac pacemaker or defibrillator
* Any severe chronic medical condition that compromises cardiac or respiratory status
* Patients with acute lower respiratory tract infections requiring antibiotic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Penetration aspiration scores on videofluoroscopy (number of swallows out of 6 that score 3 or more on the penetration aspiration scale) (Hypothesis 2 protocols 1 and 2) | 1 hour post intervention and 2 weeks post intervention
  Penetration aspiration scores on videofluoroscopy (number of swallows out of 6 that score 3 or more on the penetration aspiration scale)

SECONDARY OUTCOMES:
Improvement of: Functional oral ingestion scale (FOIS) and or the dysphagia severity rating scale (DSRS) (Hypothesis 2 protocol 2) | 2 weeks post intervention
  Improvement of: Functional oral ingestion scale (FOIS) and or the dysphagia severity rating scale (DSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, MBChB, PhD, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Upper G.I laboratory, Salford Royal Hospital, Manchester, Greater Manchester
  - Stroke Unit, Nottingham University Hospitals, Nottingham, Notthinghamshire

IPD SHARING:
Plan to Share IPD: No
No identifiable individual participant information will be shared outside the immediate research team. However, identifiable individual participant information will be made available to the Medical research council and the University of Manchester if required for the purposes of auditing the study.

REFERENCES:
- [Background] Smithard DG, O'Neill PA, Parks C, Morris J. Complications and outcome after acute stroke. Does dysphagia matter? Stroke. 1996 Jul;27(7):1200-4. doi: 10.1161/01.str.27.7.1200. PMID 8685928
- [Background] Geeganage C, Beavan J, Ellender S, Bath PM. Interventions for dysphagia and nutritional support in acute and subacute stroke. Cochrane Database Syst Rev. 2012 Oct 17;10:CD000323. doi: 10.1002/14651858.CD000323.pub2. PMID 23076886
- [Background] Finucane TE, Bynum JP. Use of tube feeding to prevent aspiration pneumonia. Lancet. 1996 Nov 23;348(9039):1421-4. doi: 10.1016/S0140-6736(96)03369-7. No abstract available. PMID 8937283
- [Background] Machado AG, Baker KB, Schuster D, Butler RS, Rezai A. Chronic electrical stimulation of the contralesional lateral cerebellar nucleus enhances recovery of motor function after cerebral ischemia in rats. Brain Res. 2009 Jul 14;1280:107-16. doi: 10.1016/j.brainres.2009.05.007. Epub 2009 May 12. PMID 19445910
- [Background] Park HJ, Furmaga H, Cooperrider J, Gale JT, Baker KB, Machado AG. Modulation of Cortical Motor Evoked Potential After Stroke During Electrical Stimulation of the Lateral Cerebellar Nucleus. Brain Stimul. 2015 Nov-Dec;8(6):1043-8. doi: 10.1016/j.brs.2015.06.020. Epub 2015 Jul 8. PMID 26215752
- [Background] Hamdy S, Rothwell JC, Brooks DJ, Bailey D, Aziz Q, Thompson DG. Identification of the cerebral loci processing human swallowing with H2(15)O PET activation. J Neurophysiol. 1999 Apr;81(4):1917-26. doi: 10.1152/jn.1999.81.4.1917. PMID 10200226
- [Background] Jayasekeran V, Rothwell J, Hamdy S. Non-invasive magnetic stimulation of the human cerebellum facilitates cortico-bulbar projections in the swallowing motor system. Neurogastroenterol Motil. 2011 Sep;23(9):831-e341. doi: 10.1111/j.1365-2982.2011.01747.x. PMID 21838728
- [Background] Vasant DH, Michou E, Mistry S, Rothwell JC, Hamdy S. High-frequency focal repetitive cerebellar stimulation induces prolonged increases in human pharyngeal motor cortex excitability. J Physiol. 2015 Nov 15;593(22):4963-77. doi: 10.1113/JP270817. Epub 2015 Sep 30. PMID 26316351
- [Background] Mistry S, Verin E, Singh S, Jefferson S, Rothwell JC, Thompson DG, Hamdy S. Unilateral suppression of pharyngeal motor cortex to repetitive transcranial magnetic stimulation reveals functional asymmetry in the hemispheric projections to human swallowing. J Physiol. 2007 Dec 1;585(Pt 2):525-38. doi: 10.1113/jphysiol.2007.144592. Epub 2007 Oct 11. PMID 17932140
- [Background] Hamdy S, Rothwell JC. Gut feelings about recovery after stroke: the organization and reorganization of human swallowing motor cortex. Trends Neurosci. 1998 Jul;21(7):278-82. doi: 10.1016/s0166-2236(97)01212-5. PMID 9683316
- [Background] Hamdy S, Aziz Q, Rothwell JC, Singh KD, Barlow J, Hughes DG, Tallis RC, Thompson DG. The cortical topography of human swallowing musculature in health and disease. Nat Med. 1996 Nov;2(11):1217-24. doi: 10.1038/nm1196-1217. PMID 8898748
- [Background] Hamdy S, Mikulis DJ, Crawley A, Xue S, Lau H, Henry S, Diamant NE. Cortical activation during human volitional swallowing: an event-related fMRI study. Am J Physiol. 1999 Jul;277(1):G219-25. doi: 10.1152/ajpgi.1999.277.1.G219. PMID 10409170
- [Background] Hamdy S, Aziz Q, Rothwell JC, Power M, Singh KD, Nicholson DA, Tallis RC, Thompson DG. Recovery of swallowing after dysphagic stroke relates to functional reorganization in the intact motor cortex. Gastroenterology. 1998 Nov;115(5):1104-12. doi: 10.1016/s0016-5085(98)70081-2. PMID 9797365
- [Background] Hamdy S, Rothwell JC, Aziz Q, Singh KD, Thompson DG. Long-term reorganization of human motor cortex driven by short-term sensory stimulation. Nat Neurosci. 1998 May;1(1):64-8. doi: 10.1038/264. PMID 10195111
- [Background] Fraser C, Power M, Hamdy S, Rothwell J, Hobday D, Hollander I, Tyrell P, Hobson A, Williams S, Thompson D. Driving plasticity in human adult motor cortex is associated with improved motor function after brain injury. Neuron. 2002 May 30;34(5):831-40. doi: 10.1016/s0896-6273(02)00705-5. PMID 12062028
- [Background] Siebner HR, Rothwell J. Transcranial magnetic stimulation: new insights into representational cortical plasticity. Exp Brain Res. 2003 Jan;148(1):1-16. doi: 10.1007/s00221-002-1234-2. Epub 2002 Nov 5. PMID 12478392
- [Background] Gow D, Rothwell J, Hobson A, Thompson D, Hamdy S. Induction of long-term plasticity in human swallowing motor cortex following repetitive cortical stimulation. Clin Neurophysiol. 2004 May;115(5):1044-51. doi: 10.1016/j.clinph.2003.12.001. PMID 15066528
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Jefferson S, Mistry S, Michou E, Singh S, Rothwell JC, Hamdy S. Reversal of a virtual lesion in human pharyngeal motor cortex by high frequency contralesional brain stimulation. Gastroenterology. 2009 Sep;137(3):841-9, 849.e1. doi: 10.1053/j.gastro.2009.04.056. Epub 2009 May 7. PMID 19427312
- [Background] Jayasekeran V, Singh S, Tyrrell P, Michou E, Jefferson S, Mistry S, Gamble E, Rothwell J, Thompson D, Hamdy S. Adjunctive functional pharyngeal electrical stimulation reverses swallowing disability after brain lesions. Gastroenterology. 2010 May;138(5):1737-46. doi: 10.1053/j.gastro.2010.01.052. Epub 2010 Feb 2. PMID 20138037
- [Background] Vasant DH, Mistry S, Michou E, Jefferson S, Rothwell JC, Hamdy S. Transcranial direct current stimulation reverses neurophysiological and behavioural effects of focal inhibition of human pharyngeal motor cortex on swallowing. J Physiol. 2014 Feb 15;592(4):695-709. doi: 10.1113/jphysiol.2013.263475. Epub 2013 Nov 18. PMID 24247983